CLINICAL TRIAL: NCT06223997
Title: Exploring the Experiences of Adults Living With Multiple Pre-existing Long-term Conditions and Long COVID to Understand Their Rehabilitation Needs
Brief Title: The Impact of Long COVID on People Living With Pre-existing LTC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0948
Record Dates: First submitted 2024-01-24; First posted 2024-01-25 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Long COVID; Multiple Chronic Conditions
Keywords: COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Multiple Chronic Conditions; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the impact of long COVID on people who have multiple (two or more) pre-existing long-term conditions (such as diabetes and asthma). The main question it aims to answer is:

• How does long COVID impact the lives of adults living with multiple pre-existing long-term conditions and what are their rehabilitation needs?

Participants will be asked to:

* Take photos of things they feel represent the impact of long COVID on their day-to-day lives across seven days and,
* Take part in an interview to discuss the impact of long COVID.

DETAILED DESCRIPTION:
This qualitative study will involve participants taking photographs (during their usual day-to-day activities), followed by 1:1 semi-structured interviews. Participants will be adults living with multiple pre-existing long-term conditions (LTC) and long COVID or their carers/supporters.

Stage 1: Photographs Participants will be asked to take photographs of things they feel represent or symbolise the impact of long COVID on their day-to-day lives across seven days in advance of the interview.

Stage 2: Interviews Semi-structured 1:1 interviews will be held face-to-face, online or telephone (in accordance with participant preference to optimise inclusivity). The iterative interview topic guide will continue to be informed by patient and public involvement and engagement, evidence (including preceding projects of the PhD), and the participants' photographs. Photographs will be viewed during the interview with participants.

The findings of this qualitative study will be used to inform the adaptation of exercise-based rehabilitation programmes to improve health and well-being which meets the needs of individuals living with multiple pre-existing LTC and long COVID.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) living with long COVID (or 'post-COVID-19 condition' in accordance with the World Health Organisation definition) and ≥2 pre-existing long-term conditions or carer/supporter for someone who is
* Living in Leicester (UK)
* Able to take photographs or carer/supporter who is able and willing
* Able and willing to provide informed consent

Exclusion Criteria:

* Child (<18 years)
* Unable to participate in a face-to-face, online or telephone interview
* Unable to access interpreter for first language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be individuals living with multiple (≥2) pre-existing long-term conditions and long COVID or 'post-COVID-19 condition' (in accordance with the World Health Organisation definition) or carer/supporter for someone who is; identified and recruited via University Hospitals of Leicester NHS Trust. Participants will be living in Leicester (UK) and either able to take photographs themselves or have a carer/supporter who is able and willing to do this for them.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Experiences and perceptions of the impact of long COVID on health and well-being | April - August 2024
  Participant photographs and 1:1 semi-structured interviews will be used to explore the experiences and perceptions of purposive samples of adults living with multiple pre-existing long-term conditions and long COVID to understand their rehabilitation needs. Photovoice and photo-elicitation will be used in combination with reflexive thematic analysis to support the interpretation process and a more participant led understanding of concepts.

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Dr Evans, Principal Investigator — University of Leicester

IPD SHARING:
Plan to Share IPD: No